CLINICAL TRIAL: NCT07296276
Title: A Prospective, Single Arm, Open-label, Interventional Study to Evaluate the Accuracy and Precision of the Continuous Glucose Monitoring System 'CareSens Air 3' in Adult Patients With Type 1 Diabetes
Brief Title: Accuracy and Precision of the Continuous Glucose Monitoring System 'CareSens Air 3' in Adult Patients With T1DM
Acronym: Air3Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: i-SENS, Inc. (Industry)
Collaborators: Integrated Medical Development (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CGM-008A-P102
Record Dates: First submitted 2025-12-11; First posted 2025-12-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Induction of low and high blood glucose.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The CareSens Air 3 data will neither be available to the investigational site nor the participants during the course of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CareSens Air 3 primary insertion site (Experimental): CareSens Air 3 primary insertion site
  Interventions: Device: CareSens Air 3 primary insertion
- CareSens Air 3 secondary insertion site (Experimental): CareSens Air 3 secondary insertion site
  Interventions: Device: CareSens Air 3 secondary insertion

INTERVENTIONS:
Device: CareSens Air 3 primary insertion — Primary CareSens Air 3 device
  Arms: CareSens Air 3 primary insertion site
Device: CareSens Air 3 secondary insertion — Secondary CareSens Air 3 device
  Arms: CareSens Air 3 secondary insertion site

SUMMARY:
This is a prospective, single arm, open-label, interventional, pilot study to evaluate the accuracy and precision of the continuous glucose monitoring (CGM) system of i-SENS, Inc., CareSens Air 3, in adult patients with type 1 diabetes.

DETAILED DESCRIPTION:
Participants will wear two CareSens Air 3 and one Libre 3 Plus for 16 days without access to glucose values from the CareSens Air 3 devices while maintaining their original diabetes mellitus treatment. The participants will draw capillary blood at least 8 times a day using the SMBG system between study visits.

Between insertion and removal of the CareSens Air 3 the participants will be in the clinic 4 times to obtain accurate glucose reading from the reference device under carefully controlled circumstances including induction of low and high blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are 18-65 years of age, inclusive
* Patients with type 1 diabetes who use intensive insulin therapy (multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII) including users of systems with continuous glucose monitoring (CGM) driven automatic adjustment of insulin doses for at least 3 months
* Patients who voluntarily decide to participate in the study and provide written informed consent

Exclusion Criteria:

* The following abnormal skin or skin diseases or skin alterations at the CGM sensor attachment or insertion site: Severe psoriasis, recent burn injury or severe sunburn, severe eczema, severe scar, extensive tattoo, dermatitis herpetiformis, severe rash, Staphylococcus aureus infection.
* Allergic contact dermatitis to medical adhesives.
* History of frequent catheter abscesses associated with pump therapy.
* Severe hypoglycemia events within 3 months prior to screening. Severe hypoglycemia is defined as loss of consciousness or seizure requiring emergency medical treatment due to hypoglycemia.
* Hypoglycemia unawareness.
* Conditions that predispose to hypoglycemia including inadequately treated thyroid and adrenal disease.
* Participants with diabetic ketoacidosis within 3 months prior to screening.
* History of epilepsy or syncope within 6 months prior to screening.
* Unstable vascular diseases (defined by event or increasing symptoms in the last 6 months) or with insufficient therapy, including: Stroke, transitory cerebral ischemia, ischemic heart disease, peripheral vascular disease, and serious arrhythmia.
* Patients with anemia (hemoglobin below normal range).
* Patients scheduled for X-ray, MRI, CT or diathermy during the study.
* Pregnant or lactating women or those who plan to become pregnant or do not agree to use an adequate method of contraception during the study.
* Patients who are currently participating or participated within 2 weeks prior to screening in another study or plan to participate in another study that in the opinion of the investigator would affect the safety of the study participant or the study result.
* Patients unwilling to abstain from ingesting the foodstuffs listed in Appendix 3 in excess of the allowed amounts.
* Patients with cognitive impairment or who are not suitable for this study or may be at increased risk associated with study participation in the opinion of the investigator.
* Wearing of a pace maker or other comparable medical devices.
* HbA1c >9.5%.
* Dependency from the sponsor or the clinical investigator.
* Unwillingness and/or inability to comply with study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the glucose concentration measurements | 16 days
  percentage of iCGM values in the measuring range less than 70 mg/dL (3.9 mmol/l) within +/- 15 mg/dL (0.83 mmol/l) of the reference venous glucose measurement by YSI analyzer

SECONDARY OUTCOMES:
Precision of the glucose measurements | 16 days
  Precision (absolute relative difference between simultaneous measurements between two CGM devices)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Headlands Research AMCR, Escondido, California
  - Diablo Clinical Research, Walnut Creek, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rainier Clinical Reseach Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No
The plan is to publish the results, but to keep the individual data proprietary.